CLINICAL TRIAL: NCT00604383
Title: Phase 3, Multicenter,Parallel,Randomized Dbl-masked,Placebo-controlled Study of the Effects of 32 mg/dy Ruboxistaurin Vision Loss in Patients With Type 1 or Type 2 Diabetes Mellitus and an Early Treatment Diabetic Retinopathy Study Level Between 47A and 53E.
Brief Title: Protein Kinase C (PKC) Inhibitor-Diabetic Retinopathy Phase 3 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4743; B7A-MC-MBCM (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ruboxistaurin (Experimental)
  Interventions: Drug: ruboxistaurin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ruboxistaurin — 32-mg tablet, orally, daily, up to 42 months
  Other Names: LY333531
  Arms: Ruboxistaurin
Drug: placebo — 1 tablet, orally, daily, up to 42 months
  Arms: Placebo

SUMMARY:
This study is to test whether or not 32 milligrams (mg) of ruboxistaurin a day over three years will reduce vision loss associated with diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* 18 years or older
* Meet specific requirements for diabetic retinopathy
* Free of severe or chronically disabling conditions, except diabetes, diabetic retinopathy and diabetic macular edema
* Hemoglobin A1c (HbA1C) ≤13.0%

Exclusion Criteria:

* History of panretinal photocoagulation for diabetic retinopathy, conditions that might affect the progression of diabetic retinopathy, or unstable angina
* Investigators, site personnel directly affiliated with the study and their families
* Presence of eye disorders that may affect the progression of diabetic retinopathy or cause vision loss
* Presence of medical disorder, cancer, or elevated laboratory measurements that could represent a safety risk during the study
* Women who are pregnant, breastfeeding, intend to become pregnant, or who are sexually active without using an acceptable method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2001-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beutner, Study Director — Chromaderm, Inc.
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT -5 hours, EST) or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Davis MD, Sheetz MJ, Aiello LP, Milton RC, Danis RP, Zhi X, Girach A, Jimenez MC, Vignati L; PKC-DRS2 Study Group. Effect of ruboxistaurin on the visual acuity decline associated with long-standing diabetic macular edema. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):1-4. doi: 10.1167/iovs.08-2473. Epub 2008 Aug 15. PMID 18708615
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 36-month treatment phase and a 0 to 6-month extended treatment phase. Completers are those who completed the 36-month treatment phase.
Groups:
- Ruboxistaurin: One 32-milligram (mg) tablet, orally, daily, for up to 42 months
- Placebo: 1 tablet, orally, daily, for up to 42 months
Period: Overall Study
Arm/Group | Ruboxistaurin | Placebo
Started | 345 | 340
Received at Least 1 Dose of Study Drug | 345 | 340
Received Extended Treatment | 136 | 141
Completed | 258 | 256
Not Completed | 87 | 84
Not completed — Withdrawal by Subject | 33 | 31
Not completed — Lost to Follow-up | 24 | 19
Not completed — Death | 14 | 22
Not completed — Adverse Event | 16 | 9
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ruboxistaurin: One 32-mg tablet, orally, daily, for up to 42 months
- Total: Total of all reporting groups
Arm/Group | Ruboxistaurin | Placebo | Total
Number analyzed (Participants) | 345 | 340 | 685
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.48 (10.91) | 59.18 (10.61) | 59.33 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 122 | 252
  Male | 215 | 218 | 433
Race/Ethnicity, Customized [Number; unit: participants]
  African Descent | 43 | 27 | 70
  Caucasian | 259 | 273 | 532
  East/Southeast Asian | 15 | 12 | 27
  Hispanic | 18 | 20 | 38
  Other | 9 | 8 | 17
  Western Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 345 | 340 | 685

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Sustained Moderate Visual Loss (SMVL) as Defined as a Visual Acuity Loss of ≥15 Letters Measured Twice During a 6-month Period
Description: SMVL is defined as a ≥15-letter decrease from baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) that the participant sustained during the last 6 months of study participation (Months 30-36). Participants who discontinued the study early may have had SMVL if there was a 6-month period of ≥15 letters lost in VA ending with the last visit at which VA was assessed. ETDRS visual acuity uses an eye chart with 5 letters per line. The scores range from 0 (no letters read correctly) to 100 (all letters read correctly). Percentage of participants = (number of participants who had SMVL) / (number of participants who were randomized) * 100.
Time Frame: Baseline through 36 months
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Ruboxistaurin: One 32-mg tablet, orally, daily, for 36 months
- Placebo: 1 tablet, orally, daily, for 36 months
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 345 | 340
percentage of participants | 5.5 | 9.1
Statistical Analysis 1: Comparison: Ruboxistaurin vs Placebo; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants Who Developed Center Involved or Imminently Threatened Diabetic Macular Edema (DME)
Description: DME is the accumulation of extracellular fluid in the retinal tissue of the macular area, which can reduce the ability for fine visual discrimination. Percentage of participants = (number of participants who developed center involved or imminently threatened DME) / (number of participants who had no center involved or imminently threatened DME at baseline) * 100.
Time Frame: Baseline through 36 months
Population: All randomized participants who had no center involved or imminently threatened DME at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 248 | 249
percentage of participants | 44.4 | 49.0

3. Secondary Outcome: Percentage of Participants Who Experienced the Development of Proliferative Diabetic Retinopathy (PDR)
Description: Percentage of participants = (number of participants who experienced the development of PDR) / (number of participants who were randomized) * 100.
Time Frame: Baseline through 36 months
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 345 | 340
percentage of participants | 35.9 | 36.5

4. Secondary Outcome: Change From Baseline up to 36 Months in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25)
Description: NEI-VFQ-25 consisted of 25 questions and was used to measure the influence of visual disability and symptoms on general health of participants. The possible total score range for the NEI-VFQ-25 was from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: Baseline, up to 36 months
Population: All randomized participants with evaluable NEI-VFQ-25 total score. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 290 | 289
units on a scale | -3.82 (14.75) | -4.10 (13.45)

5. Secondary Outcome: Change From Baseline up to 36 Months in Mental and Physical Components of the Medical Outcomes Study 36-Item Short Form (SF-36) Health Status Questionnaire
Description: SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions. There are 2 component scores, mental component score (MCS) and physical component score (PCS). MCS score consisted of social functioning, vitality, mental health, and role-emotional scales. PCS score consisted of physical functioning, bodily pain, role-physical, and general health scales. Both MCS and PCS have scores ranging from 0 to 100 with higher scores indicating better mental or physical health.
Time Frame: Baseline, up to 36 months
Population: All randomized participants with evaluable SF-36 MCS and PCS. LOCF was used to impute missing post-baseline values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ruboxistaurin | Placebo
Number analyzed (Participants) | 290 | 289
units on a scale
  MCS | -12.21 (70.91) | -19.85 (70.05)
  PCS | -30.63 (84.92) | -29.15 (79.41)

ADVERSE EVENTS:
Arm/Group | Ruboxistaurin | Placebo
Serious Adverse Events (participants affected / at risk) | 145/345 | 157/340
Other Adverse Events (participants affected / at risk) | 314/345 | 322/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ruboxistaurin (N=345) | Placebo (N=340)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 13 (13)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 6 (6)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 5 (6) | 4 (4)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 11 (11)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 25 (38) | 19 (26)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery atherosclerosis (Cardiac disorders) | 1 (1) | 1 (2)
Coronary artery disease (Cardiac disorders) | 30 (38) | 30 (33)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 3 (3)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 13 (16)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (3) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular neuronitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (3)
Retinal detachment (Eye disorders) | 0 (0) | 4 (4)
Retinal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (3)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 2 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (2)
Colonic haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 10 (12) | 4 (4)
Death (General disorders) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 5 (6)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 5 (5)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertensive gastropathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 3 (3)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis acute (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 12 (16) | 12 (13)
Clostridium colitis (Infections and infestations) | 4 (4) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 3 (4)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 2 (2)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 2 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 8 (9) | 6 (9)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (15) | 13 (15)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative infection (Infections and infestations) | 1 (1) | 3 (3)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 4 (4)
Septic embolus (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 2 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 4 (5)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Closed head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Coagulation time abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 7 (9)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Lower limb deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/130 (0) | 1/122 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/215 (0) | 1/218 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 8 (9)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 4 (5) | 7 (8)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (2) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 6 (6)
Renal failure acute (Renal and urinary disorders) | 14 (18) | 12 (12)
Renal failure chronic (Renal and urinary disorders) | 9 (12) | 5 (6)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/215 (1) | 0/218 (0)
Priapism (Reproductive system and breast disorders) | 0/215 (0) | 1/218 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (7)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 3 (4)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 7 (8) | 8 (9)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypoperfusion (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 3 (4) | 3 (4)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 3 (3)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruboxistaurin (N=345) | Placebo (N=340)
Anaemia (Blood and lymphatic system disorders) | 30 (33) | 36 (37)
Dry eye (Eye disorders) | 17 (19) | 19 (21)
Eye pain (Eye disorders) | 22 (30) | 18 (28)
Maculopathy (Eye disorders) | 14 (19) | 17 (17)
Vision blurred (Eye disorders) | 18 (22) | 19 (26)
Visual disturbance (Eye disorders) | 19 (26) | 20 (26)
Vitreous floaters (Eye disorders) | 19 (26) | 15 (17)
Vitreous haemorrhage (Eye disorders) | 17 (20) | 20 (24)
Constipation (Gastrointestinal disorders) | 21 (24) | 21 (22)
Diarrhoea (Gastrointestinal disorders) | 32 (37) | 40 (104)
Dyspepsia (Gastrointestinal disorders) | 19 (22) | 12 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 27 (27) | 21 (21)
Nausea (Gastrointestinal disorders) | 26 (33) | 37 (46)
Vomiting (Gastrointestinal disorders) | 20 (24) | 33 (56)
Asthenia (General disorders) | 18 (30) | 17 (19)
Chest pain (General disorders) | 17 (24) | 22 (32)
Fatigue (General disorders) | 19 (23) | 19 (21)
Oedema peripheral (General disorders) | 61 (73) | 67 (99)
Pyrexia (General disorders) | 19 (26) | 16 (20)
Bronchitis (Infections and infestations) | 24 (30) | 29 (38)
Influenza (Infections and infestations) | 44 (55) | 45 (49)
Localised infection (Infections and infestations) | 21 (29) | 22 (29)
Nasopharyngitis (Infections and infestations) | 59 (91) | 67 (112)
Onychomycosis (Infections and infestations) | 18 (19) | 18 (19)
Pneumonia (Infections and infestations) | 11 (12) | 17 (19)
Sinusitis (Infections and infestations) | 25 (38) | 32 (43)
Upper respiratory tract infection (Infections and infestations) | 23 (29) | 35 (51)
Urinary tract infection (Infections and infestations) | 25 (33) | 31 (44)
Contusion (Injury, poisoning and procedural complications) | 12 (19) | 23 (26)
Fall (Injury, poisoning and procedural complications) | 18 (19) | 17 (23)
Blood cholesterol increased (Investigations) | 25 (25) | 16 (16)
Cardiac murmur (Investigations) | 26 (26) | 21 (22)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 30 (30) | 28 (28)
Obesity (Metabolism and nutrition disorders) | 14 (14) | 18 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 36 (44)
Arthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 20 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (36) | 27 (34)
Joint swelling (Musculoskeletal and connective tissue disorders) | 27 (32) | 29 (39)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (16) | 18 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (44) | 35 (50)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 18 (23) | 13 (15)
Dizziness (Nervous system disorders) | 29 (40) | 27 (30)
Headache (Nervous system disorders) | 33 (39) | 45 (59)
Hypoaesthesia (Nervous system disorders) | 21 (23) | 33 (36)
Neuropathy peripheral (Nervous system disorders) | 19 (21) | 15 (15)
Anxiety (Psychiatric disorders) | 13 (13) | 18 (22)
Depression (Psychiatric disorders) | 28 (28) | 31 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 57 (78) | 42 (60)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (35) | 30 (33)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (28) | 29 (35)
Skin ulcer (Skin and subcutaneous tissue disorders) | 21 (25) | 21 (28)
Hypertension (Vascular disorders) | 58 (58) | 50 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days